CLINICAL TRIAL: NCT05945316
Title: Performance Improvement: Does Mock Code Simulation Improve the Confidence Level of Newly Graduated Nurses?
Status: Completed | Type: Observational
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 008.NUR.2022.C
Record Dates: First submitted 2023-07-06; First posted 2023-07-14 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Mock Code Training Simulation

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Behavioral: Accessing Confidence levels of Nursing students — Three mock CODE BLUE training events for Spring, Summer, and Fall Nursing Residents and Nursing Fellows are scheduled for 2022 followed by an actively participated CODE BLUE event. The PI plan to collect data from all new residents meeting the inclusion/exclusion criteria with voluntary participation to complete.
  Other Names: Performance during CODE BLUE over time

SUMMARY:
The study is a descriptive correlational study over three surveys that will examine the improvement of confidence level associated between the implementation of mock code training simulation and the real live event.

DETAILED DESCRIPTION:
Participants will be asked to respond online to a questionnaire or survey launched via Survey Monkey®. Demographic information will be collected first Appendix B. A self-reported confidence level via the Student Satisfaction and self-confidence in learning scale will be utilized and serves as a data collection tool. The scale will be deployed via email as a scale A B and C Appendix C to each study participant and is the same scale. The participants will complete survey A after completion of the initial educational simulation training the survey B will be completed when the participants attended an unannounced simulation activity. Survey C will be completed after the first actively involved Code Blue situation. The survey is a 13-item instrument designed to measure student satisfaction five items with the simulation activity and self-confidence in learning eight items using a five-point scale. Reliability was tested using Cronbach's alpha: satisfaction equals 0.94 self-confidence equals 0.87 Franklin Burns and Lee 2014.

ELIGIBILITY:
Inclusion Criteria:

All newly graduated nurses and nurse fellows in a residency training program at MCMC Able to read and understand English

Exclusion Criteria:

Clinical staff not affiliated with the residency and fellowship program.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All newly graduated nurses and nurse fellows in a residency training program at MCMC Able to read and understand English
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2022-03-16 (Actual); Primary Completion 2025-07-22 (Actual); Study Completion 2025-07-22 (Actual)

PRIMARY OUTCOMES:
Accessing Confidence levels of Nursing students during CODE BLUE | 2 years
  The confidence level will be measured utilizing the Student Satisfaction and Self-Confidence in Learning Scale (SCLS). SCLS is a 13-item survey instrument designed to measure student satisfaction (five items) with the simulation activity and self-confidence in learning (eight items). Statements will be confirmed with answers on a five-point Likert scale: strongly disagree (1), disagree (2), undecided (3), agree (4), and strongly agree (5). Measures will occur during three different activities.

SECONDARY OUTCOMES:
Simulated cardiopulmonary resuscitation will improve confidence level in newly graduated nurses and nurse fellows during their residency training | 2 yrs
  The confidence level will be measured utilizing the Student Satisfaction and Self Confidence in Learning Scale (SCLS). SCLS is a 13-item survey instrument designed to measure student satisfaction (five items) with the simulation activity and self-confidence in learning (eight items). Statements will be confirmed with answers on a five-point Likert scale: strongly disagree (1), disagree (2), undecided (3), agree (4), and strongly agree (5). Measures will occur during three different activities.

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Gret Friedrich-Cuntz, EdD, Principal Investigator — Methodist Charlton Medical Center (Methodist Health System-
Locations (1):
- Methodist Dallas Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
The PI is committed to disseminate research results in a timely fashion. Sharing of results generated by the data analysis during the course of the project will be through presentation at national scientific meetings and/or publication in open access journals. All information obtained will be source de-identified and presented on a large scale and not traceable to any one particular individual.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will become available with in 1 to 2 years. All study-related documents will be retained by the CRI until at least three years after study completion or according to local laws, whichever is longer. . Records will also be accessible to MHS staff upon request unless constituting a violation of patient confidentiality.
Access Criteria: All study-related documents will be retained by the CRI until at least three years after study completion or according to local laws, whichever is longer. . Records will also be accessible to MHS staff upon request unless constituting a violation of patient confidentiality.

REFERENCES:
- [Background] Advice, P.R.N. (2004). Staff development: Mock code, real value. Nursing2004
- [Background] Carroll L, Pignataro S. Use of portable simulation manikins to increase the frequency of mock code training on four inpatient surgical units. J Contin Educ Nurs. 2009 Jun;40(6):250-1. doi: 10.3928/00220124-20090522-04. PMID 19639913
- [Background] Carney P. Mock code: a game that saves lives. RN (For Managers). 1983 Jul;46(7):18P. No abstract available. PMID 6553335
- [Background] Cardoza MP, Hood PA. Comparative study of baccalaureate nursing student self-efficacy before and after simulation. Comput Inform Nurs. 2012 Mar;30(3):142-7. doi: 10.1097/NCN.0b013e3182388936. PMID 22080746
- [Background] Franklin AE, Burns P, Lee CS. Psychometric testing on the NLN Student Satisfaction and Self-Confidence in Learning, Simulation Design Scale, and Educational Practices Questionnaire using a sample of pre-licensure novice nurses. Nurse Educ Today. 2014 Oct;34(10):1298-304. doi: 10.1016/j.nedt.2014.06.011. Epub 2014 Jul 9. PMID 25066650
- [Background] Hill CR, Dickter L, Van Daalen EM. A matter of life and death: the implementation of a Mock Code Blue Program in acute care. Medsurg Nurs. 2010 Sep-Oct;19(5):300-2, 304. No abstract available. PMID 21189744
- [Background] Huseman KF. Improving code blue response through the use of simulation. J Nurses Staff Dev. 2012 May-Jun;28(3):120-4. doi: 10.1097/NND.0b013e3182551506. PMID 22617782
- [Background] Kakora-Shiner N. Using ward-based simulation in cardiopulmonary training. Nurs Stand. 2009 May 27-Jun 2;23(38):42-7. doi: 10.7748/ns2009.05.23.38.42.c6975. PMID 19552045
- [Background] Marsch SC, Muller C, Marquardt K, Conrad G, Tschan F, Hunziker PR. Human factors affect the quality of cardiopulmonary resuscitation in simulated cardiac arrests. Resuscitation. 2004 Jan;60(1):51-6. doi: 10.1016/j.resuscitation.2003.08.004. PMID 14987784
- [Background] Ngo DQ, Vu C, Nguyen T, Sotolongo P, Talati M, Zahabi N, Platt K. The Effect of Mock Code Blue Simulations and Dedicated Advanced Cardiac Life Support Didactics on Resident Perceived Competency. Cureus. 2020 Nov 25;12(11):e11705. doi: 10.7759/cureus.11705. PMID 33391938